CLINICAL TRIAL: NCT03101787
Title: Early Initiation of Extracorporeal Life Support in Refractory OHCA (INCEPTION)
Brief Title: Early Initiation of Extracorporeal Life Support in Refractory OHCA
Acronym: INCEPTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Getinge Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL58067.068.16
Record Dates: First submitted 2017-03-30; First posted 2017-04-05 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-08

CONDITIONS: Cardiac Arrest; Out-Of-Hospital Cardiac Arrest; Sudden Cardiac Death
Keywords: ECPR; Extracorporeal CardioPulmonary Resuscitation; OHCA; Out-of-Hospital Cardiac Arrest; CPR; CardioPulmonary Resuscitation; ECMO; ExtraCorporeal Membrane Oxygenation; Refractory Cardiac Arrest
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest; Death, Sudden, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CCPR protocol (No Intervention): Preclinical Cardiopulmonary resuscitation (CPR) by emergency medical services (EMS) and rapid transport to the emergency department with ongoing mechanical CPR and advanced cardiac life support (ACLS).
  Clinical Upon the patient's arrival, the standard of care (CCPR) will be continued according to ERC guidelines.
  No special preparations for the trial are needed before the patient's arrival.
- ECPR protocol (Experimental): Preclinical Cardiopulmonary resuscitation (CPR) by emergency medical services (EMS) and transport to the emergency department with ongoing mechanical CPR and advanced cardiac life support (ACLS).
  Clinical The ECPR team is mobilized while the patient is transported to the hospital. Initiation of extracorporeal cardiopulmonary resuscitation (ECPR).
  Time from arrest to start of cannulation is < 60 minutes.
  Interventions: Procedure: Extracorporeal cardiopulmonary resuscitation (ECPR)

INTERVENTIONS:
Procedure: Extracorporeal cardiopulmonary resuscitation (ECPR) — In addition to the routine response team, the ECLS team are called to the ED while the patient is transported to the hospital.
  The team consists of a physician skilled and qualified in femoral cannulation, a perfusionist and a scrub nurse.
  Upon the patient's arrival at the emergency department, CPR will be continued, with continuation of mechanical chest compressions with minimization of interruptions.
  Time from arrest to start of cannulation is < 60 minutes.
  Arms: ECPR protocol

SUMMARY:
Despite adequate conventional cardiopulmonary resuscitation (CCPR) and attempted defibrillation, a considerable number of patients in cardiac arrest fail to achieve sustained return of spontaneous circulation. The INCEPTION trial is a multicenter, randomized controlled trial that will explore extracorporeal cardiopulmonary resuscitation (ECPR) in patients in refractory out-of-hospital cardiac arrest (OHCA) presenting with ventricular fibrillation or tachycardia. It aims to determine the effect on survival and neurological outcome. Additionally, it will evaluate the feasibility and cost-effectiveness of ECPR.

DETAILED DESCRIPTION:
There are approximately 275,000 cases of out-of-hospital cardiac arrest (OHCA) per year in Europe, of which two-thirds have a primary cardiac origin. However, despite adequate conventional cardiopulmonary resuscitation (CCPR) and attempted defibrillation, a considerable number of these patients fail to achieve sustained return of spontaneous circulation (ROSC).

Treatment of the underlying cause of the arrest, in most cases coronary artery occlusion, is paramount. But in the absence of ROSC, the possibilities to perform these life-saving interventions are limited. Continued CCPR is currently the standard of care for these patients. Initiation of extracorporeal cardiopulmonary resuscitation (ECPR) restores circulation, with the potential to minimize (or even reversing) organ damage, prevent re-arrest due to ischemia-triggered myocardial dysfunction and providing a bridge to possible diagnosis and treatment. Several studies have demonstrated that ECPR is feasible and may be advantageous with respect to survival and neurological outcome.

The INCEPTION trial aims to compare ECPR to CCPR in the population that is expected to benefit the most from this intervention: young patients presenting with ventricular fibrillation or tachycardia (VF/VT) and a refractory cardiac arrest. Furthermore, it will provide data on the cost-effectiveness of this intervention, which to date has been unavailable. Although the costs may prove to be high, the gain in quality-adjusted life years (QALY's) may be substantial given the fact that most patients are relatively young and the current alternative carries a poor prognosis. This can determine whether ECPR should be pursued as a standard of care in patients with refractory arrest.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 - ≤70 years
2. Witnessed OHCA (by bystanders)
3. Initial rhythm of VF/VT or AED administered
4. Bystander BLS

Exclusion Criteria:

1. ROSC within 15 minutes of conventional CPR with sustained hemodynamic recovery
2. Terminal heart failure (NYHA III or IV)
3. Severe pulmonary disease (COPD GIII of GIV)
4. Disseminated oncological disease
5. Obvious or suspected pregnancy
6. Bilateral femoral bypass surgery
7. Known contraindications for ECPR
8. Known pre-arrest CPC-score of 3 or 4
9. Known limitations in therapy or a Do Not Resuscitate-order
10. Multitrauma (Injury Severity Score >15)
11. Expected time-to-start cannulation > 60 minutes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
30-day survival rate with favorable neurological status | 30 days
  Favorable neurological status is defined as 1 or 2 on the using Cerebral Performance Category scale

SECONDARY OUTCOMES:
Neurological outcome on the CPC scale | 30 days, 3 months, 6 months and 12 months
  Does ECPR improve the neurological outcome at 30 days, 3 months, 6 months and 12 months on the CPC scale
Quality Adjusted Life Years (QALY's) | 30 days, 3 months, 6 months and 12 months
  Does ECPR improve the amount of Quality Adjusted Life Years (QALY's) at 30 days, 3 months, 6 months and 12 months
Reason for discontinuation of treatment between the treatment groups | Within 1 year
  Is there a difference in reason for discontinuation of treatment between the treatment groups
Time to return of circulation | Within 1 year
  What is the time to return of circulation
Additional costs of ECPR with respect to CCPR | 1 year
  What are the additional costs of ECPR with respect to CCPR
Costs per gained QALY for ECPR vs. CCPR | 1 year
  What are the costs per gained QALY for ECPR vs. CCPR
Length of stay at the ICU | 1 year
  Is there a difference in length of stay at the ICU between the treatment groups
Length of stay at the hospital | 1 year
  Is there a difference in length of stay at the hospital between the treatment groups
Duration of clinical rehabilitation time | 1 year
  Is there a difference in the duration of clinical rehabilitation time
Duration of mechanical ventilation | 1 year
  Is there a difference in the duration of mechanical ventilation between treatment groups
Need for renal replacement therapy | 1 year
  Is there a difference in need for renal replacement therapy between the treatment groups
Acute kidney injury according to the RIFLE criteria | 1 year
  Is there a difference in acute kidney injury according to the RIFLE criteria
Time to target hypothermia | 1 year
  Is there a difference in time to target hypothermia between the treatment groups
Difference in metabolic markers between treatment groups | 6 days
  Is there a difference in metabolic markers such as (1) pH, (2) etCO2, (3) ScVO2 and (4) lactate at arrival at the ED, right after initialization of circulation (either by ROSC or ECPR), 1, 2, 3, 4, 5 and 6 hours after return of circulation and at 1, 2, 3, 4, 5 and 6 days after the OHCA between the treatment groups
Difference in metabolic markers between between the survivors and non-survivors | 6 days
  Is there a difference in metabolic markers such as (1) pH, (2) etCO2, (3) ScVO2 and (4) lactate at arrival at the ED, right after initialization of circulation (either by ROSC or ECPR), 1, 2, 3, 4, 5 and 6 hours after return of circulation and at 1, 2, 3, 4, 5 and 6 days after the OHCA between the survivors and non-survivors

CONTACTS AND LOCATIONS:
Overall Officials: Marcel van de Poll, MD, PhD, Principal Investigator — Maastricht UMC
Locations (10):
- Netherlands (10):
  - Maastricht UMC, Maastricht, Limburg
  - Catharina Ziekenhuis, Eindhoven, North Brabant
  - Academisch Medisch Centrum, Amsterdam, North Holland
  - Isala Klinieken, Zwolle, Overijssel
  - Leids Universitair Medisch Centrum, Leiden, South Holland
  - St. Antonius Hospital, Nieuwegein, Utrecht
  - Onze Lieve Vrouwen Gasthuis, Amsterdam
  - Erasmus MC, Rotterdam
  - HagaZiekenhuis, The Hague
  - Universitair Medisch Centrum Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Verberght HCR, Delnoij TSR, Suverein MM, Lunsing J, Hermanides RC, Otterspoor L, Elzo Kraemer CV, Vlaar APJ, van der Heijden JJ, Scholten E, Uil CAD, Miranda DDR, Akin S, Metz J, van der Horst ICC, Mathot BJ, de Jonge J, Nijboer MWN, de Meijer VE, Sanders JSF, Christiaans MHL, van Zuilen AD, Hagenaars H, Wind J, Danhof M, Olde Damink SWM, Winkens B, Maessen JG, Lorusso R, van de Poll MCG; INCEPTION-investigators. Organ Donor Potential After Extracorporeal Cardiopulmonary Resuscitation for Out-of-Hospital Cardiac Arrest: A Post-Hoc Analysis of a Randomized Controlled Trial. Clin Transplant. 2025 Nov;39(11):e70382. doi: 10.1111/ctr.70382. PMID 41243868
- [Derived] Ubben JFH, Heuts S, Delnoij TSR, Suverein MM, Hermanides RC, Otterspoor LC, Kraemer CVE, Vlaar APJ, van der Heijden JJ, Scholten E, den Uil C, Dos Reis Miranda D, Akin S, de Metz J, van der Horst ICC, Winkens B, Maessen JG, Lorusso R, van de Poll MCG. Favorable resuscitation characteristics in patients undergoing extracorporeal cardiopulmonary resuscitation: A secondary analysis of the INCEPTION-trial. Resusc Plus. 2024 May 13;18:100657. doi: 10.1016/j.resplu.2024.100657. eCollection 2024 Jun. PMID 38778803
- [Derived] Heuts S, van de Koolwijk AF, Gabrio A, Ubben JFH, van der Horst ICC, Delnoij TSR, Suverein MM, Maessen JG, Lorusso R, van de Poll MCG. Extracorporeal life support in cardiac arrest: a post hoc Bayesian re-analysis of the INCEPTION trial. Eur Heart J Acute Cardiovasc Care. 2024 Feb 16;13(2):191-200. doi: 10.1093/ehjacc/zuad130. PMID 37872725
- [Derived] Suverein MM, Delnoij TSR, Lorusso R, Brandon Bravo Bruinsma GJ, Otterspoor L, Elzo Kraemer CV, Vlaar APJ, van der Heijden JJ, Scholten E, den Uil C, Jansen T, van den Bogaard B, Kuijpers M, Lam KY, Montero Cabezas JM, Driessen AHG, Rittersma SZH, Heijnen BG, Dos Reis Miranda D, Bleeker G, de Metz J, Hermanides RS, Lopez Matta J, Eberl S, Donker DW, van Thiel RJ, Akin S, van Meer O, Henriques J, Bokhoven KC, Mandigers L, Bunge JJH, Bol ME, Winkens B, Essers B, Weerwind PW, Maessen JG, van de Poll MCG. Early Extracorporeal CPR for Refractory Out-of-Hospital Cardiac Arrest. N Engl J Med. 2023 Jan 26;388(4):299-309. doi: 10.1056/NEJMoa2204511. PMID 36720132
- [Derived] Bol ME, Suverein MM, Lorusso R, Delnoij TSR, Brandon Bravo Bruinsma GJ, Otterspoor L, Kuijpers M, Lam KY, Vlaar APJ, Elzo Kraemer CV, van der Heijden JJ, Scholten E, Driessen AHG, Montero Cabezas JM, Rittersma SZH, Heijnen BG, Taccone FS, Essers B, Delhaas T, Weerwind PW, Roekaerts PMHJ, Maessen JG, van de Poll MCG. Early initiation of extracorporeal life support in refractory out-of-hospital cardiac arrest: Design and rationale of the INCEPTION trial. Am Heart J. 2019 Apr;210:58-68. doi: 10.1016/j.ahj.2018.12.008. Epub 2018 Dec 14. PMID 30738245